CLINICAL TRIAL: NCT07193940
Title: Flexible Ureteroscopy Versus Extracorporeal Shock Wave Lithotripsy for Treatment of Lower Calyceal Renal Stones Less Than 15 mm: A Prospective Randomized Comparative Study
Brief Title: Flexible Ureteroscopy Versus Extracorporeal Shock Wave Lithotripsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Mohamed Abdellatif, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ureteroscopy VS ESWL
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi | interventions — Lithotripsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Ureteroscopy (Experimental): Interventional procedure: Flexible Ureteroscopy
  Interventions: Procedure: Flexible Ureteroscopy
- Extracorporeal Shock Wave Lithotripsy (Experimental): Extracorporeal Shock Wave Lithotripsy (ESWL)
  Interventions: Procedure: extracorporeal shock wave lithotripsy (ESWL)

INTERVENTIONS:
Procedure: Flexible Ureteroscopy — Flexible Ureterorenoscopy
  Arms: Flexible Ureteroscopy
Procedure: extracorporeal shock wave lithotripsy (ESWL) — extracorporeal shock wave lithotripsy (ESWL)
  Arms: Extracorporeal Shock Wave Lithotripsy

SUMMARY:
To compare the efficacy and safety of flexible ureterorenoscopy (fURS) versus extracorporeal shock wave lithotripsy (ESWL) in managing lower calyceal renal stones ≤15 mm and <1000 HU.

DETAILED DESCRIPTION:
Urolithiasis is a common condition with a steadily increasing global prevalence, and lower calyceal stone treatment is particularly challenging. While stones ≤15 mm and <1000 Hounsfield Units (HU) are generally treatable, lower pole anatomy limits fragment clearance after extracorporeal shock wave lithotripsy (ESWL). Published SFR for ESWL in this location range between 60-80%, which are lower compared to other calyceal sites. Predictive factors such as stone density, size, and skin-to-stone distance are applied to optimize patients selection.

Conversely, flexible ureteroscopy (fURS) with laser lithotripsy achieves more and higher quality SFRs (80-95%) by active fragmentation and retrieval of the stones, thereby bypassing the anatomic barriers. However, It is invasive, requires anesthesia and has complications such as ureteral trauma and infection, including a small but certain risk of sepsis. EAU and AUA guidelines currently recommend either ESWL or URS for stones <20 mm, but note reduced clearance of lower-pole stones by ESWL.

This creates a therapeutic dilemma: should stones ≤15 mm and <1000 HU, theoretically ideal for ESWL, nevertheless to be managed non-invasively, or should fURS be given priority because of increased reliability? We anticipate that fURS will provide a higher 3-month stone-free rate than ESWL, though ESWL may remain a suitable first-line treatment in well-selected patients owing to lower morbidity and non-invasive nature.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 y)
* Lower-calyx stone
* Less than or equal15 mm
* Mean Hounsfield (HU) <1000

Exclusion Criteria:

* Pregnancy
* Uncorrected coagulopathy
* Active UTI/obstruction
* Anatomical barriers to Flexible Ureteroscopy or extracorporeal shock wave lithotripsy coupling (e.g., prohibitive SSD/BMI).
* Cardiac devices contraindicating ESWL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate at 1 months on low-dose NCCT (no fragment >2 mm; report CIRF separately) | baseline
  Stone-free rate at 1 months on low-dose NCCT (no fragment >2 mm; report CIRF separately)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

REFERENCES:
- [Result] Ng CF. The effect of stone size, location, and number on the outcome of extracorporeal shock wave lithotripsy. Int Braz J Urol. 2008;34(6):759-66. Available from: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2684300/
- [Result] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Result] Sampaio FJ, Aragao AH. Inferior pole collecting system anatomy: its probable role in extracorporeal shock wave lithotripsy. J Urol. 1992 Feb;147(2):322-4. doi: 10.1016/s0022-5347(17)37226-9. PMID 1732584
- [Result] Akman T, Binbay M, Ozgor F, Ugurlu M, Tekinarslan E, Kezer C, Aslan R, Muslumanoglu AY. Comparison of percutaneous nephrolithotomy and retrograde flexible nephrolithotripsy for the management of 2-4 cm stones: a matched-pair analysis. BJU Int. 2012 May;109(9):1384-9. doi: 10.1111/j.1464-410X.2011.10691.x. Epub 2011 Oct 28. PMID 22093679
- [Result] Somani BK, Giusti G, Sun Y, Osther PJ, Frank M, De Sio M, Turna B, de la Rosette J. Complications associated with ureterorenoscopy (URS) related to treatment of urolithiasis: the Clinical Research Office of Endourological Society URS Global study. World J Urol. 2017 Apr;35(4):675-681. doi: 10.1007/s00345-016-1909-0. Epub 2016 Aug 4. PMID 27492012
- [Result] Fankhauser CD, Weber D, Muntener M, Poyet C, Sulser T, Hermanns T. Effectiveness of Flexible Ureterorenoscopy Versus Extracorporeal Shock Wave Lithotripsy for Renal Calculi of 5-15 mm: Results of a Randomized Controlled Trial. Eur Urol Open Sci. 2021 Feb 2;25:5-10. doi: 10.1016/j.euros.2021.01.001. eCollection 2021 Mar. PMID 34337498
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2684300/